CLINICAL TRIAL: NCT03272555
Title: WILD 5 Wellness: A 30-Day Intervention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failed study, participants showed no improvements
Sponsor: Beloit College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 365
Record Dates: First submitted 2017-08-29; First posted 2017-09-05 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Wellness; Anxiety; Depression; Cognitive and Executive Dysfunction
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Participants (Other): The participants in this arm will engage in the WILD 5 Wellness activities combining five wellness elements including exercise, mindfulness, sleep, social connectedness and nutrition.
  Interventions: Other: WILD 5 Wellness Interventions

INTERVENTIONS:
Other: WILD 5 Wellness Interventions — Students enrolled in the study will be asked to complete activities in five wellness elements including exercise, mindfulness, sleep, social connectedness and nutrition for 30 days.

SUMMARY:
The purpose of this study is to explore the efficacy and feasibility of an integrated, prescriptive, and trackable wellness intervention combining five wellness elements including exercise, mindfulness, sleep, social connectedness, and nutrition in First Year Beloit College students self-selected into a wellness focused first year initiative.

DETAILED DESCRIPTION:
The purpose of this study is to explore the efficacy and feasibility of an integrated, prescriptive, and trackable wellness intervention combining five wellness elements including exercise, mindfulness, sleep, social connectedness, and nutrition in First Year Beloit College students self-selected into a wellness focused first year initiative. This program is called "WILD 5 Wellness: A 30-Day Intervention". Results for this study will be quantified through the use of standardized self-report questionnaires administered prior to and after students complete the WILD 5 program. Data will be collected to evaluate participants' adherence and response to each element of WILD 5, a 5-pronged 30-day wellness intervention. It is expected that this 30-day integrated, prescriptive, and trackable program will be found to be an efficacious wellness intervention for First Year Beloit College students.

ELIGIBILITY:
Inclusion Criteria:

* students 18 years of age or older
* students enrolled in First Year Initiative Course titled, "Habits of Mind, Habits of Body."

Exclusion Criteria:

* individuals who are pregnant or plan to get pregnant during the next 30 days
* students who are not enrolled in the First Year Initiative Course titled, "Habits of Mind, Habits of Body".

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-13 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) | Day 0, Day 31+/- 5 days, Day 30+6 months (approximately)
  PHQ-9 is a self reported depression scale.
Change in Generalized Anxiety Disorder-7 (GAD-7) | Day 0, Day 31+/- 5 days, Day 30+6 months (approximately)
  GAD-7 is a self-reported questionnaire used to assess anxiety symptoms.
Change in The HERO Wellness Scale | Day 0, Day 31+/- 5 days, Day 30+6 months (approximately)
  The HERO Wellness Scale is a brief scale designed to measure mental wellness specifically happiness, enthusiasm, resilience and optimism.
Change in World Health Organization-5 (WHO-5) | Day 0, Day 31+/- 5 days, Day 30+6 months (approximately)
  WHO-5 is a brief scale that measures mental well-bring.
Change in Cognitive and Physical Functioning Questionnaire (CPFQ) | Day 0, Day 31+/- 5 days, Day 30+6 months (approximately)
  CPFQ is a brief scale that measures cognitive and executive dysfunction.

SECONDARY OUTCOMES:
The Post-Program Participant Questionnaire | Day 31+/- 5 days
  The Post-Program Participant Questionnaire is a brief survey that captures participants' opinions about WILD 5 Wellness: A 30-Day Intervention, and subjective ranking of their overall wellness.

CONTACTS AND LOCATIONS:
Locations (1):
- Beloit College, Beloit, Wisconsin, United States